CLINICAL TRIAL: NCT06647472
Title: Proteomic Analysis on Myopic Children Using Orthokeratology Lenses With Good or Poor Myopic Control. The ProMOC Study
Brief Title: Proteomic Analysis on Myopic Children Using Orthokeratology Lenses With Good or Poor Myopic Control
Acronym: ProMOC
Status: Active, not recruiting | Type: Observational
Sponsor: Vejle Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: The ProMOC study
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Myopia; Healthy; Orthokeratology
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The key objective of the study is to gain an understanding of the biochemical processes that contribute to orthokeratology lenses being more effective in specific individuals compared to others. With this knowledge, we hope to optimize treatment effectiveness in those currently experiencing less favorable outcomes from treatment in the future.

The primary aim is to investigate differences in protein levels in children using orthokeratology lenses with various effects of myopia control.

Hypothesis: There is a significant difference in the expression of molecules in children with various effects of myopia control.

ELIGIBILITY:
Inclusion Criteria:

* Children treated with orthokeratology lenses.
* Children on or above the 95th percentile of myopia growth curves for European children at the time of treatment initiation.
* Treatment and follow-up duration ≥ 6 months.

Exclusion Criteria:

* Current use of eye drops.
* Objective signs of dry eyes on slit-lamp examination.
* Active eye infection.

Ages: 5 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: Children who are currently being treated with orthokeratology lenses at the Ophthalmic Department, Vejle Hospital, University Hospital of Southern Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Difference in protein levels measured by mass spectrometry label-free quantification (LFQ) between children using orthokeratology lenses with different levels of myopia control effectiveness | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Øjenafdelingen, Vejle Sygehus, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-03-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT06647472/SAP_000.pdf